CLINICAL TRIAL: NCT03157362
Title: Effects of Social Presence and Perception in Virtual Reality on Pain
Acronym: SPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1701006910
Record Dates: First submitted 2017-05-09; First posted 2017-05-17 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Chronic Pain, Widespread
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Each participant will experience four conditions, in a random order, crossing "near" and "far" virtual environments, and social presence or no social presence.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be informed of what condition they are assigned to. The research assistants who code the data will also not be informed of condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Time 1 (Active Comparator): Participant will be randomly assigned to one of the four interventions; either Near Non-Social, Near Social, Far Non-Social, or Far Social
  Interventions: Other: Near Non-Social; Other: Near Social; Other: Far Non-Social; Other: Far Social
- Time 2 (Active Comparator): Participant will be randomly assigned to one of the remaining three interventions; either Near Non-Social, Near Social, Far Non-Social, or Far Social
  Interventions: Other: Near Non-Social; Other: Near Social; Other: Far Non-Social; Other: Far Social
- Time 3 (Active Comparator): Participant will be randomly assigned to one of the remaining two interventions; either Near Non-Social, Near Social, Far Non-Social, or Far Social
  Interventions: Other: Near Non-Social; Other: Near Social; Other: Far Non-Social; Other: Far Social
- Time 4 (Active Comparator): Participant will complete the remaining intervention; either Near Non-Social, Near Social, Far Non-Social, or Far Social
  Interventions: Other: Near Non-Social; Other: Near Social; Other: Far Non-Social; Other: Far Social

INTERVENTIONS:
Other: Near Non-Social — Participants will be stably seated, and observed by a research assistant, as they complete an induced pain threshold task while they experience a virtual environment that reproduces the room in which they are seated.
Other: Near Social — Participants will be stably seated, and observed by a research assistant, as they complete an induced pain threshold task while they experience a virtual environment that reproduces the room in which they are seated, and converse with a confederate represented by an avatar.
Other: Far Non-Social — Participants will be stably seated, and observed by a research assistant, as they complete an induced pain threshold task while they experience a virtual environment that reproduces a different room.
Other: Far Social — Participants will be stably seated, and observed by a research assistant, as they complete an induced pain threshold task while they experience a virtual environment that reproduces another room, and converse with a confederate represented by an avatar.

SUMMARY:
This experiment aims to examine the effects of transportation via social presence in "near" and "far" virtual environments, on pain threshold in two groups: 1. healthy volunteers in an induced pain task, and 2. older adults suffering from pain. In the first, pilot group, a within-subjects study, participants will complete a series of induced-pain heat ramps in virtual environments that are "near" or "far"-in other words, they will either duplicate their actual physical environment, or represent another location. A second factor in this experiment will be mediated social presence, in which participants interact with confederates as avatars in either condition. The hypotheses follow: H1: Participants who feel present in a remote location will have a higher pain tolerance than those in a near location. H2: Participants who feel socially present with a confederate will have a higher pain tolerance than those who are alone in a virtual environment. H3: There will be an interaction between social presence and virtual environment such that participants who feel socially present in a remote location will have the highest pain tolerance overall. Building on these results,the next step will be a long-term study on older adult pain patients. In this step, the most successful condition in the first study to lightweight, portable headsets that can be used outside of the lab environment. This intervention will be tested on older adult patients who are suffering from chronic pain.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE: Virtual reality (VR) has been used to treat pain for over 15 years but the mechanism of pain relief remains to be fully explored. Virtual reality is a particularly high-presence medium, in that people using VR tend to react to mediated content as if it were salient to their physical selves. Like this sense of presence, pain is a subjective phenomenon- it exists only as perceived by an individual. The vivid and interactive nature of VR creates a sense of presence in the virtual world, or in virtual bodies, by plausibly replacing sensory information from the real world with sensory information that creates a virtual environment and/or body. Previous work has found that presence in virtual environments reduces pain. Presence in virtual reality, and in media in general, is frequently referred to metaphorically as transportation. For example, people say about someone who's reading a book, "She's in another world" or complain, "he's not present with me now, he's distracted by your phone." When a person in pain subjectively feels that he or she is not present in the real-world location of the painful stimulus, his or her sense of actual or potential damage may be less, and therefore his or her pain tolerance may be greater. One component of virtual worlds that may affect pain perception is thus their ability to "transport" the viewer to locations other than the hospital, their home, or other places where they are experiencing pain. Previous pilot work on presence in remote environments in virtual reality indicated that presence in a "far" as opposed to a "near" virtual environment increased pain tolerance in an induced pain task. While these results point towards the idea that transportation through presence in virtual reality can increase pain tolerance or increase pain threshold, this result requires more support to justify deploying to a patient population. However, virtual worlds also allow for social interaction, which has the potential to strongly affect both pain and the sensation of presence in an environment. While social support has been linked to pain reduction, in a recent study, participants who texted with a stranger while undergoing surgery were less likely to require analgesia than those who texted with companions or played a distracting game on their phone. While the authors propose that the context of the chat may have affected participants' pain levels, another additive possibility is that these patients were experiencing social presence with the strangers, who were conversing from a location outside the hospital, and were thus feeling less present in the hospital environment. This might explain why participants received greater benefit from these text conversations than from conversations with loved ones, who were conversing from the hospital environment where their pain occurred. This aligns with other research that shows that participants in a text conversation estimate the physical distance to their conversational partner to be greater if they feel less socially present with that conversational partner. The following experiment will compare the effects of social presence and transportation in immersive virtual reality environments, and serve as a baseline to design more widely accessible interventions.

METHODS AND RESEARCH STRATEGY: A power analysis on a between-subjects pilot study on normal participants comparing near and far virtual environments suggests 48.5 participants for a power of .8. This study is a within-subjects design which should require less power. However, to account for participant attrition 75 participants will be invited to the first pilot study. In order to rapidly collect this number of patients with minimal risk, data collection will begin with a student sample of convenience. The most successful stimuli will then be modified to trial in older adults in a long-term study looking at VR for patients already suffering from pain. In the first sample, participants will visit the lab once to complete an experiment lasting less than one hour. Each participant will experience four conditions crossing "near" and "far" virtual environments, and social presence or no social presence. (In this experiment, social presence will be operationalized as a conversation with a confederate represented by an avatar). Participants will be stably seated, and observed by a research assistant, as they experience four environments: 1. A virtual environment that reproduces the room in which they are seated. 2. A virtual environment that reproduces the room in which they are seated, in which participants will view and converse with a confederate represented by an avatar. 3. Another location. 4. Another location, in which participants will view and converse with a confederate represented by an avatar. Confederates will follow a script to keep the conversations of similar length and content. During each condition, participants will complete an induced pain task using a Medoc TSA-2001/Model Q-Sense thermode. (For more detailed discussion of this device, and of the stimulus justification, please see the Human Subjects Issues section of the Data Safety Monitoring Plan). Prior to experiencing the four experimental conditions, participants will complete a "practice" induced pain task while viewing a duplication of the virtual environment. This will allow them to orient themselves to both the virtual environment and the pain task, since based on the pilot experiment, order effects are predicted to be most notable for the first pain task administered. In this and all subsequent induced pain tasks, participants will place their non-dominant hand on the thermode and will be instructed to remove their hand as soon as they feel the temperature has become "painful". The beginning and end of each trial (when the heat ramp begins, and when participants remove their hands) will be noted, and that time duration, and thus the degree of temperature to which it corresponds, will serve as the measure of pain threshold for that trial. In addition to this outcome measure, after each pain trial participants will also fill out a brief self-report survey. These measures will include their self-reported feelings of presence in the virtual environment, and social presence with the confederate. The survey will also include manipulation checks to establish whether participants believed the confederate to be a real person, and whether they believed that the confederate was in the location described in each condition. All subsequent conditions will be presented in a randomized order to control for order effects, and conducted as follows. The time to complete these surveys will be approximately 7-10 minutes, which will also allow participants time between each trial to reorient themselves to the real environment, and for any lingering effects of heat on their hands to dissipate. Finally, participants' movements will be tracked in order to provide an additional indication of how participants engaged with the virtual environment.

ELIGIBILITY:
Inclusion Criteria:

Consenting adult

Exclusion Criteria:

1. History of cardiovascular disorder
2. History of fainting or seizures
3. Open cut or sore on hand to be thermally tested
4. Burn or sunburn on hand to be thermally tested.
5. Pregnancy
6. Prone to motion sickness, or have balance or dizziness conditions
7. Recent concussion
8. Seizure disorders
9. History of fainting or seizures
10. Visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Pain threshold in degrees tolerated at end of trial | The beginning and end of each trial < 90 seconds
  Change in temperature from the beginning to the end of each trial (when the heat ramp begins, and when participants remove their hands) will be noted in milliseconds.

SECONDARY OUTCOMES:
Self-reported social presence | ~15 minutes at the end of each trial
  Questionnaire of self-reported feelings of social presence with the confederate
Self-reported environmental presence | ~15 minutes at the end of each trial
  Questionnaire of self-reported feelings of presence in the virtual environment

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell Virtual Embodiment Lab, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffman HG, Doctor JN, Patterson DR, Carrougher GJ, Furness TA 3rd. Virtual reality as an adjunctive pain control during burn wound care in adolescent patients. Pain. 2000 Mar;85(1-2):305-9. doi: 10.1016/s0304-3959(99)00275-4. PMID 10692634
- [Background] F. P. Brooks Jr, 1990. Virtual reality at work. Human Machine Interfaces for Teleoperators and Virtual Environments, 67.
- [Background] Moseley GL. A pain neuromatrix approach to patients with chronic pain. Man Ther. 2003 Aug;8(3):130-40. doi: 10.1016/s1356-689x(03)00051-1. PMID 12909433
- [Background] Sanchez-Vives MV, Slater M. From presence to consciousness through virtual reality. Nat Rev Neurosci. 2005 Apr;6(4):332-9. doi: 10.1038/nrn1651. PMID 15803164
- [Background] Hoffman HG, Sharar SR, Coda B, Everett JJ, Ciol M, Richards T, Patterson DR. Manipulating presence influences the magnitude of virtual reality analgesia. Pain. 2004 Sep;111(1-2):162-8. doi: 10.1016/j.pain.2004.06.013. PMID 15327820
- [Background] de Tommaso M, Ricci K, Laneve L, Savino N, Antonaci V, Livrea P. Virtual visual effect of hospital waiting room on pain modulation in healthy subjects and patients with chronic migraine. Pain Res Treat. 2013;2013:515730. doi: 10.1155/2013/515730. Epub 2013 Jan 10. PMID 23365736
- [Background] Brown JL, Sheffield D, Leary MR, Robinson ME. Social support and experimental pain. Psychosom Med. 2003 Mar-Apr;65(2):276-83. doi: 10.1097/01.psy.0000030388.62434.46. PMID 12651995
- [Background] Guillory JE, Hancock JT, Woodruff C, Keilman J. Text messaging reduces analgesic requirements during surgery. Pain Med. 2015 Apr;16(4):667-72. doi: 10.1111/pme.12610. Epub 2014 Dec 19. PMID 25529995